CLINICAL TRIAL: NCT06393595
Title: Prediction of Outcomes in Patients With Chronic Heart Failure Based on Tissue Raman Spectroscopy
Acronym: PROMETHEUS
Status: Completed | Type: Observational
Sponsor: Samara State Medical University (Other)
Collaborators: City Clinical Hospital No.1 named after N.I. Pirogov (Other)
Responsible Party: Sponsor
Other Study IDs: CHF-RS001
Record Dates: First submitted 2024-04-26; First posted 2024-05-01 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Chronic Heart Failure
Keywords: cumulative death; cardiovascular death (CVD); CVD or hospitalization for heart failure exacerbation; surface enhanced Raman Spectroscopy; skin Raman Spectroscopy
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 2 ml of blood serum from each participant for Raman spectroscopy were collected and processed. All other biochemical analysis were provided by hospital central laboratory
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CHD + CHF: Coronary Heart Disease with overt Chronic Heart Failure (200 participants)
  Interventions: Diagnostic Test: surface enhanced Raman Spectroscopy
- CHD: Coronary Heart Disease without Chronic Heart Failure (70 participants)
  Interventions: Diagnostic Test: surface enhanced Raman Spectroscopy
- NICMP +CHF: Non-Ischemic Cardiomyopathies with overt Chronic Heart Failure (50 participants)
  Interventions: Diagnostic Test: surface enhanced Raman Spectroscopy
- VCMP+CHF: Valvular Cardiomyopathies with overt Chronic Heart Failure (40 participants)
  Interventions: Diagnostic Test: surface enhanced Raman Spectroscopy

INTERVENTIONS:
Diagnostic Test: surface enhanced Raman Spectroscopy — Spectral measurements of blood serum were performed on a silver nanoparticle substrate. Each 1.5 μL serum sample was applied to a substrate with a layer of silver nanoparticles and dried . The spectral characteristics of serum were analyzed using an experimental bench consisting of a spectrometric system and a microscope . The spectra were excited by laser module with a center wavelength of 785 nm. Each of the obtained spectra was a discrete set of 1700 parameters .
  For skin Raman spectroscopy an experimental portable RS system was used, including a 785 nm diode laser , a portable commercially available Raman probe to filter the collected scattered radiation, and a portable spectrometer (QE65Pro, Ocean optics, Florida, USA). The scattered radiation was collected from the upper 1 to 2 mm thick skin layer. The Raman spectral range was 780-1000 nm with resolution of 0.2 nm. Each spectrum was recorded at an exposure time of 20 seconds with three-fold accumulation.
  Other Names: Skin Raman Spectroscopy

SUMMARY:
Chronic heart failure (CHF) is a syndrome complicating heart disease, the prevalence of which has reached epidemic levels. According to global statistics the most common causes of CHF are coronary heart disease (CHD): 26.5%, arterial hypertension (AH):26.2% . The category of patients with CHD complicated by CHF prevails in clinical practice, requiring an optimized approach to determining prognosis in order to improve the effectiveness of therapy. In the literature, this issue has been studied with the use of general clinical, biochemical, instrumental criteria. Nevertheless, the problem of optimized prognosis in patients with CHF remains. Its solution may lie in the study of metabolic parameters of biological media - skin, blood serum by Raman spectroscopy.

Skin is an accessible tissue for studying the effects of a wide range of age-dependent noncommunicable diseases, including cardiovascular disease, type 2 diabetes mellitus, and chronic kidney disease. We were one of the first to use skin RS as a method of determining renal dysfunction, a necessary component of chronic kidney disease. However, the applicability of RS/SERS in the diagnosis and prognosis of specific diseases, as well as in the collection of statistical data for this analytical approach, remains an open question . Despite the fact that the method is classified as analytical, it can be used to identify not so much specific chemical molecules as their specific loci, which provide vibrations that change the wavelengths of the scattered spectrum. The resulting spectrum can be presented as a metabolic "portrait" of the disease, with the most informative loci, the combination of which is associated with a negative prognosis.

The innovative analytical methods of optical spectroscopy proposed in this project provide new level information about hundreds of molecules and their active centers that have prospects as biomarkers. This study aims to determine the clinical relevance of skin and serum RS in patients with CHF, realized on state-of-the-art instrumentation in a comprehensive patient study setting. The research proposed in this project will contribute to the development of high-tech production of new optical devices for rapid diagnosis and prognosis of a wide range of diseases.

DETAILED DESCRIPTION:
This study included participants hospitalized in the cardiology unit of Samara city Clinical Hospital No.1 n.a. N.I.Pirogov of Emergency Medical Aid.The reason for hospitalization was newly diagnosed chronic heart failure or its exacerbation.

Objective: 1) to develop a personalized approach to prediction of total mortality, cardiovascular death in patients with CHD complicated by CHF on the basis of Raman spectra of skin, plasma, blood serum.

2)To develop a classification of Raman spectra characteristic for CHF, as well as its phenotypes and relevant comorbid conditions - Chronic kidney disease (CKD) and glycemic status.

Study Material:

1. Group with CHF based on CHD of both sexes aged 35 to 84 years (200 participants);
2. Group with CHD without CHF (70 participants);
3. Group with CHF with non-ischemic cardiomyopathies (50 participants);
4. group with CHF and valvular cardiomyopathies (40 participants)

The study design is divided into two consecutive parts:

A)cross-sectional cohort . B)prospective

Cross-sectional study (part 1). Material: groups 1-4.

Objectives:

1. To identify Raman spectral characteristics specific to the CHF syndrome, skin RS and serum SERS would be performed in groups of different CHF etiology: noncomplicated CHD ; CHD complicated by CHF; non-ischemic Cardiomyopathies (CMP) complicated by CHF(Dilated CMP, Inflammatory CMP,; valvular CMPs ).
2. To study the influence of CHF phenotypes (divided by Left Ventricular ejection fraction (LVEF)), as well as comorbidity - chronic kidney disease, type 2 diabetes mellitus(DM2) on skin and serum Raman spectra, biochemical parameters in the group with CHD.

   Prospective study (part 2) Study material: group 1.

   Objectives:
3. To establish the possibilities of serum SERS and skin RS parameters in predicting overall mortality in patients with CHD complicated by CHF in comparison with prediction models based on parameters of clinical, biochemical and instrumental routine techniques.
4. Develop prediction models for total mortality, CV mortality, and CV mortality in combination with hospitalizations for CHD participants with CHF .
5. To establish relationships with the most prognostically important spectral components of RS and known markers of atherosclerosis and cardiovascular diseases (CVD): CKD parameters; troponin T, glucose; cholesterol spectrum parameters.

Planned period of the cross-sectional phase of the study: November 2022 to May 2023.

Visit 1- Determination of inclusion/exclusion criteria for recruitment. Collection of clinical, biochemical, instrumental parameters. Determination of serum SERS and skin RS.

Planned period of the prospective study: November 2022-May 2024. Visit -1 is used to include only participants from group (1) in the prospective part of the study: CHD+CHF.

Visit-2 is planned at 4-6 months after the initial evaluation. The aim of visit-to assess patient's clinical status and compliance to prescribed medication.

Visit 3 (end of prospective follow-up ).The purpose of the visit - to collect information about hospitalizations and complications that occurred after visit 2. In case of death according to relatives' information, to confirm the fact of death in the electronic medical information analytical system (EMIAS).

Scientific novelty of the research: The technology of surface enhanced Raman spectroscopy (SERS) of blood serum on nanosilver substrate will be tested. Artificial intelligence technology is used for discriminative analysis based on SERS parameters.

Spectral features due to the influence of CVD, diabetes mellitus and renal dysfunction will be specified on RS of skin and serum SERS highlighted for the first time .

For the first time, the RS of skin, serum of non-ischemic CMPs and valvular CMPs is studied.

For the first time, a prognostic model using skin RS, SERS of patients with CHD complicated by CHF is proposed.

Based on the results of the study, models will be developed to predict mortality and cardiovascular complications in patients with CHD complicated by CHF.

Expected Results:

Mathematical models will be developed to predict cumulative mortality, CV mortality and cumulative target, including CV mortality and hospitalizations for exacerbations of CHF, based on independent predictors of biochemical, clinical, skin and serum Raman spectrometry parameters.

Spectral regions reflecting the influence of chronic heart failure syndrome as such will be identified (by comparing serum SERS of patients with different etiologies of CHF).

Spectral characteristics of three phenotypes of CHF will be identified: with preserved LVEF; moderately reduced LVEF; low LVEF.

Spectral characteristics specific for chronic kidney disease and DM2 will be identified.

ELIGIBILITY:
Inclusion Criteria:

Group 1(CHD+CHF): clinically evident CHF II-IV NYHA Classes,confirmed by NT-proBNP diagnostic levels. Any form of Coronary Heart Disease :angina pectoris up to and including 2 functional class, previous myocardial infarction, percutaneous coronary intervention or coronary arteries bypass grafts. possible functional insufficiency of A-V valves, arterial hypertension, possibly with chronic atrial fibrillation/atrial fibrillation of any form, ventricular extrasystoles of any class, Hiss bundle branch block not requiring implantation of devices, ability to self-care.

Group 2(CHD): Any form of Cronic Heart Disease :angina pectoris up to and including 2 functional class, previous myocardial infarction, percutaneous coronary intervention or coronary arteries bypass grafts, possible functional insufficiency of A-V valves of 1 stage, arterial hypertension, possibly with chronic atrial fibrillation/ flatter of any form, ventricular extrasystoles of any class, Hiss bundle branch block not requiring implantation of devices, ability to self-care.

Group 3 (NICMPs+CHF): clinically evident CHF II-IV NYHA Classes,confirmed by NT-proBNP diagnostic levels without signs of CHD in the history, without violation of coronary anatomy - stenoses (MSCT and coronary angiography). Possible functional insufficiency of A-B valves of the 1st degree, arterial hypertension, possible chronic forms of atrial fibrillation/ flatter, ventricular extrasystoles of any class, blockade of the Hiss legs not requiring implantation of devices, capable of self-care.

Group 4 (VCMPs+CHF):Valvular acquared cardiomyopathies with clinically evident CHF II-IV NYHA Classes,confirmed by NT-proBNP diagnostic levels without signs of CHD in the history, without violation of coronary anatomy - stenoses (MSCT and coronary angiography). Possible functional insufficiency of A-B valves of the 1st degree, arterial hypertension, possible chronic forms of atrial fibrillation/ flatter, ventricular extrasystoles of any class, blockade of the Hiss legs not requiring implantation of devices, capable of self-care.

Exclusion Criteria:Exclusion criteria (for groups 1-4): Acute myocardial infarction or unstable angina within the last 6 months, Dementia, lack of signed consent, CKD 4st or higher, tuberculosis, active cancer, liver cirrhosis of infectious etiology, chronic anemia : Hemoglobin less than 95 g/L, inability to self-care, type 1 diabetes mellitus,or insulin-dependent type 2 DM , anticipated heart valve surgery within one year, uncontrolled endocrine disease or malignancy likely to affect prognosis.

Ages: 35 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The researchers included participants from among those hospitalized in the cardiology department of an urban acute care hospital (groups 1,3,4)because of first-diagnosed chronic heart failure or its exacerbation.
  Group 2 consisted of patients with clinically and instrumentally proven chronic ischemic heart disease without manifestations of CHF also hospitalized. Reasons for hospitalization in this group were related to BP elevation, paroxysms of atrial fibrillation/atrial flutter.
  Selection into the study was made among consecutively admitted patients, provided that the inclusion criteria were met
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
record in electronic medical information analitical system(EMIAS) | 01.11.2022-01.05.2024
  The initial information of participant's death would be verified by official record
record in electronic medical information analitical system (EMIAS) | 01/11/2022-01/05/2024
  The initial information of participant's cardiovascular death would be verified by official record

SECONDARY OUTCOMES:
record in electronic medical information analitical system (EMIAS) and history of disease | 01/11/2022-01/05/2024
  The initial information of participant's cardiovascular death would be verified by official record . The fact of admittance to hospitals was verified by appropriate documents

OTHER OUTCOMES:
Raman spectrum classification | 11/05/2023-20/06/2024
  model of Raman spectral bands associated with chronic heart failure, LVEF, CKD,DM2

CONTACTS AND LOCATIONS:
Overall Officials: Petr A Lebedev, professor, Principal Investigator — chief of therapy chair of professional education department
Locations (1):
- city Samara hospital n.a. N.I.Pirogov, Samara, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Khristoforova YA, Bratchenko LA, Skuratova MA, Lebedeva EA, Lebedev PA, Bratchenko IA. Raman spectroscopy in chronic heart failure diagnosis based on human skin analysis. J Biophotonics. 2023 Jul;16(7):e202300016. doi: 10.1002/jbio.202300016. — https://pubmed.ncbi.nlm.nih.gov/36999197/
- See also: Konovalova DY, Lebedev PA, Zakharov VP. Raman spectroscopy of human skin for kidney failure detection. J Biophotonics. 2021 Feb;14(2):e202000360. doi: 10.1002/jbio.202000360. — https://pubmed.ncbi.nlm.nih.gov/33131189/